CLINICAL TRIAL: NCT05851703
Title: The Effects Of Instrument-Supported Cervical Manual Therapy Methods And Proprioceptive Neuromuscular Facilitation Techniques
Brief Title: The Effects Of Instrument Cervical Manual Therapy Methods And Proprioceptive Neuromuscular Facilitation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, İsmet Yurdsever, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: neck pain
Record Dates: First submitted 2023-04-30; First posted 2023-05-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Neck Pain
Keywords: pain
MeSH Terms: conditions — Neck Pain; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy applications: (Experimental): In lower cervical lateral flexion problems, pushing technique will be applied with instrument support from the articular pillar part of the superior vertebra on the side where the limitation is present
  Interventions: Other: Manual therapy application
- Proprioceptive Neuromuscular Facilitation (Experimental): Proprioceptive Neuromuscular Facilitation (PNF) techniques will be applied to the second group.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: Manual therapy application — In lower cervical lateral flexion problems, pushing technique will be applied with instrument support from the articular pillar part of the superior vertebra on the side where the limitation is present.
  In lower cervical lateral flexion problems, instrument-assisted pushing technique will be applied from the articular pillar part of the superior vertebra on the side where the limitation is present.
  Arms: Manual therapy applications:
Other: Proprioceptive Neuromuscular Facilitation — With the rhythmic initiation technique, it is to teach the movement to the person, to improve the feeling of movement, coordination and to help relaxation. With rhythmic initiation, we want the patient's initial passive and then active participation to understand the movement, the direction and rhythm of the movement. After people actively participate, they can use active joint movement.
  Arms: Proprioceptive Neuromuscular Facilitation

SUMMARY:
The location of neck pain is usually shown as "pain occurring between the occiput and the third thoracic vertebra". The annual incidence of mechanical neck pain is 12/1000 patients and is one of the most common reasons for visiting physicians. Neck pain usually lasts longer than 3 months and results in a high cost to society

DETAILED DESCRIPTION:
Movement in one plane in the cervical spine is due to the contribution of vertebrae from other planes. This complicates the kinematics and injury mechanism of the cervical region. Considering the mechanism of injury, demographic information to be obtained from the person is very important.

ELIGIBILITY:
Inclusion Criteria:

* Those with neck pain
* Being between 20-60 years old

Exclusion Criteria:

* High blood pressure
* Cardiopulmonary disease
* Malignant
* Operation, injection, etc. for the neck in the last 3 months. those with a history of treatment
* Spine surgery
* Psychological disturbance
* Neurological and orthopedic deficits

Ages: 18 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | one day
  The Neck Disability Index (NDI) measures acute and chronic neck pain or disability due to neck injury. It is the most common assessment tool used in the neck. It consists of 10 items. These; intensity of pain, personal care, lifting, reading, headaches, concentration, work, driving, sleep and leisure activities. There are 6 options in each item and the patient will mark one of these options and be evaluated accordingly.
Visual Analogue Scale | one day
  In the measurement of neck pain severity, it was planned to use a standard, proven 10 mm VAS. The severity of pain felt by the patient; It is a scale used to mark 0 = no pain and 10 = the most severe pain, thus determining the patient's pain intensity subjectively.
Algometer | one day
  It can be used to measure the sensitivity of tissues. The pressure is gradually increased and people must report the feeling of pressure applied. It has been shown that pressure algometry is a highly valid and reliable measurement of cranio-cervical muscles.
Pinchmeter | one day
  It will be used to assess finger grip strengths. Measurements will be evaluated on both hands. Before the measurements, the participants will be informed verbally and they will be allowed to experiment. When the participants are ready, they are asked to squeeze the dynamometer with all their strength for 3 seconds and then release it. Participants will rest for 1 minute between measurements.
Jamar Hand Dynomometer | one day
  The patients were placed in the sitting position with the wrist in 90° flexion and the forearm in the neutral position. Before the measurements, the participants will be informed verbally. Participants will then be asked to squeeze with all their strength for 3 seconds and then release. Participants will rest for 1 minute between measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Ismet Yurtdsever, Istanbul, None Selected, Turkey (Türkiye)

REFERENCES:
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164